CLINICAL TRIAL: NCT01881698
Title: Multiple Electrode Aggregometry and Platelet Function in Pregnancy
Brief Title: Evaluation of Platelet Function in Pregnancy With Multiple Electrode Aggregometry
Acronym: MULPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Reinhard Hahn, Principal Investigator, Medical University of Vienna
Other Study IDs: 1426/2013
Record Dates: First submitted 2013-05-17; First posted 2013-06-20 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Platelet Function; Pregnancy
Keywords: pregnancy; platelet function; monitoring; multiple electrode aggregometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Platelet function during pregnancy Multiple Electrode Aggregometry (Multiplate@) device — Observation of platelet function in pregnancy

SUMMARY:
Establishment of a range of normal values in pregnancy with the Multiple Electrode Aggregometry (Multiplate@) device, a device that allows measurement of not only platelet count but platelet function. This has not been studied in ths special patient group. Results from this trial will be used as a basis for further investigation of abnormal platelet function in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy

Exclusion Criteria:

* Rejection of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant patients above the age of majority
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Change of platelet function | 4x, as specified below
  Measurement of change of platelet function by the Multiplate® device. First measurement (baseline measurement) at enrollment into the trial. Second measurement during government-mandated gynaecological evaluation, around the 20th week of pregnancy.
  Third measurement immediately prior to delivery. Last measurement one week after delivery. 2nd, 3rd and 4th measurement for assessment of change from baseline.

SECONDARY OUTCOMES:
Platelet-associated complications | 4x, as specified below (baseline, 20th week)
  Record of bleeding events, preeclampsia, HELLP (hemolysis, elevated liver enzymes, and low platelet count) syndrome.
  Time points: at every assessment of primary outcome measure, as described above.

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Hahn, MD, Principal Investigator — Department of Anaesthesia, General Intensive Care and Pain Management, Medical University Vienna
Locations (1):
- Universitätsklinik für Frauenheilkunde, Allgemeines Krankenhaus der Stadt Wien, Vienna, Vienna, Austria